CLINICAL TRIAL: NCT02398006
Title: Figure-of-eight Bandage Versus Arm Sling for Treating Middle Third Clavicle Fractures in Adults: Study Protocol for a Randomised Controlled Trial
Brief Title: Conservative Interventions for Treating Clavicle Fractures in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Mario Lenza, Dr, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HIAE orthopaedics
Record Dates: First submitted 2015-03-12; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Fracture of Clavicle
Keywords: Clavicle [mh]; Fracture Healing [mh]; Fractures, Bone [mh]; Treatment outcome [mh]; Conservative treatment [tw]
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: a standard arm sling (Active Comparator): Group 1: the orthopaedic surgeon will apply a standard arm sling that will be used for four weeks; however, during these weeks, participants will be encouraged to discard the sling when their pain has subsided. After four weeks the same orientations of group 1 will be done to this group.
  Interventions: Other: a standard arm sling
- Group 2: a figure-of-eight bandage (Active Comparator): Group 2: a figure-of-eight bandage will be used for four weeks, and every week the participants will return to check and adjust the immobilisation. In this way, the dominant hand can remain free and simple activities will be allowed (writing, keyboarding and other). After four weeks, participants will be encouraged to discard the bandage, but load bearing will not be allowed before osseous consolidation (around 10 weeks).
  Interventions: Other: a figure-of-eight bandage

INTERVENTIONS:
Other: a standard arm sling — Closed reduction (re-aligning the fragments of the fracture) will be not performed because the reduced position is practically impossible to maintain.
  Arms: Group 1: a standard arm sling
Other: a figure-of-eight bandage — Closed reduction (re-aligning the fragments of the fracture) will be not performed because the reduced position is practically impossible to maintain.
  Arms: Group 2: a figure-of-eight bandage

SUMMARY:
Background: Fracture of the clavicle is common accounting for 2.6% to 4 % of all fractures, with an overall incidence of 36.5 to 64 per 100,000 per year. Around 80% of clavicle fractures occur in the middle third of the clavicle. There is a lack of evidence of randomised controlled trials assessing the best treatment of these fractures. The objective of this study is to evaluate the effects (benefits and harms) of conservative interventions: figure-of-eight bandage versus sling for the treating middle third clavicle fractures. Methods/Design: this project has been designed as a single-centre, parallel-group randomised controlled trial that will compare figure-of-eight bandage versus sling. The investigators aim to recruit 110 adults, aged 18 years or older, with an acute (less than 10 days) middle third clavicle fracture. Primary outcomes will be function or disability measured by DASH questionnaire; the secondary outcomes will be: modified UCLA score pain, treatment failure, adverse events and numbers returning to previous activities. Data analysis: the chi-square test will be used to analyse the results of categorical variables, and Student t-test will be used to compare groups with respect to the numerical variables. The Student t-test is used to compare the clinical outcome of each group at 1, 2 and 4 weeks and at 6 and 12 months after the intervention. The significance level of 5% (alpha = 0.05) is used for all statistical tests such that tests have a value of less than 0.05 are considered statistically significant. Discussion: According to current evidence there is very limited evidence from two single trials only regarding the effectiveness of different methods of conservative interventions for treating clavicle fractures. This study is one of the first randomised controlled trials following the CONSORT statements designed to compare two conservative methods for treating clavicle fractures (figure-of-eight versus sling).

DETAILED DESCRIPTION:
Whilst there are several options for conservative treatment for middle third clavicle fractures, only two randomised controlled published in the 80s attempted to determine the effects of different methods for conservative treatment for middle third clavicle fractures. Thus, a pragmatic trial design has been chosen as it can directly inform clinical practice; our inclusion criteria will reflect the variety in patient presentations that would be encountered by general orthopaedic surgeons in the clinical setting. The current trial includes design characteristics known to minimise bias. Participants will be assigned using a concealed random procedure, assessments and data analysis will be blinded and we will use the intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older and 65 years or less with middle third clavicle fracture,
* Acute fracture (less than 10 days), we will include all types of middle third clavicle fractures (non-displaced and displaced fractures),
* No medical contraindication to proposed methods of immobilisation,
* Understanding of Portuguese language and written informed consent.

Exclusion Criteria:

* Pathological fracture,
* Open fracture,
* Neurovascular injury on physical examination,
* Associated head injury (Glasgow Coma Scale score of <12),
* Ipsilateral upper limb fractures and/or dislocation(except hand and fingers),
* History of frozen shoulder,
* Previous disease in the limb that could influence the results (e.g. rheumatoid arthritis),
* Inability to comply with follow-up (inability to read or complete forms).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Function or disability will be measured by DASH - Disability of the Arm, Shoulder, and Hand questionnaire | 12 months
  Function or disability will be measured by DASH - Disability of the Arm, Shoulder, and Hand questionnaire validated and translated into Portuguese in Brazil, the final score of the DASH questionnaire will be converted to a percentage via the following formula: Scoring = [Sum of answers n/n - 1] X 25, where n is the number of complete answers. The two optional modules will not be measured. The value obtained will be directly proportional to the percentage of impairment of the limb function.

SECONDARY OUTCOMES:
Modified University of California at Los Angeles (modified - UCLA) | 12 months
  Modified University of California at Los Angeles (modified - UCLA), validated and translated into Portuguese in Brazil.
Pain measured on a 0 to 100 using visual analogue scale (VAS) | 12 months
  Pain measured on a 0 to 100 using visual analogue scale (VAS) (with 0 indicating no pain and 100 indicating the maximum pain). As reported in the literature, a clinically important change will be considered as a 30% or more change in pain score.
Treatment failure measured by the number of participants who have undergone or are being considered a surgical intervention | 12 months
  Treatment failure measured by the number of participants who have undergone or are being considered a surgical intervention (e.g. symptomatic non-union or malunion with intractable pain). Although studies evaluating patients with fractures without displacement reported low rates of nonunion (about 0.03%), studies with patients with displaced fractures found nonunion rates of up to 15%. Therefore, we expect between 5 and 10% of our participants might provide symptomatic nonunion during follow-up. Patients who experience this complication during follow-up study will be treated surgically with open reduction and internal fixation with pre-contoured locking plate counted down the superior surface of the clavicle and bone grafting when necessary.
Adverse events | 12 months
  Adverse events measured by: a) Cosmetic result: perception of deformity or asymmetric result (dichotomous data); b) Asymptomatic non-union (i.e. the fracture has not healed radiographically with no pain); c) Stiffness/restricted of range of shoulder movement (compared with contralateral side).
Numbers returning to previous activities (work, sport, activities of daily living), including time to return. | 12 months
  Numbers returning to previous activities (work, sport, activities of daily living), including time to return.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lenza, PhD, Principal Investigator — Hospital Israelita Albert Einstein

REFERENCES:
- [Derived] Lenza M, Taniguchi LF, Ferretti M. Figure-of-eight bandage versus arm sling for treating middle-third clavicle fractures in adults: study protocol for a randomised controlled trial. Trials. 2016 May 4;17(1):229. doi: 10.1186/s13063-016-1355-8. PMID 27142768